CLINICAL TRIAL: NCT01702129
Title: A Phase I Study of Doxorubicin-loaded Anti-EGFR Immunoliposomes in Patients With Advanced Solid Tumors
Brief Title: Anti-EGFR Immunoliposomes in Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC1
Record Dates: First submitted 2012-10-01; First posted 2012-10-05 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Solid Tumors
Keywords: EGFR; liposomes; immunoliposomes
MeSH Terms: interventions — Doxorubicin; liposomal doxorubicin; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- anti-EGFR Immunoliposomes (Experimental): anti-EGFR immunoliposomes loaded with doxorubicin. Dose escalating study. 3 patients per dose level. Dose levels: 5, 10, 20, 30, 40, 50 and 60 mg doxorubicin/m2.
  Interventions: Drug: anti-EGFR immunoliposomes loaded with doxorubicin

INTERVENTIONS:
Drug: anti-EGFR immunoliposomes loaded with doxorubicin — All patients were treated with anti-EGFR immunoliposomes Different dose levels (5, 10, 20, 30, 40, 50 and 60 mg doxorubicin/m2), at least 3 patients per dose level, treatment was given every 4 weeks
  Other Names: Doxil; cetuximab

SUMMARY:
Background: Site-specific delivery of anti-cancer therapeutics is paramount for both reducing nonspecific toxicities and increasing efficacy of chemotherapeutic agents. Due to their small molecular size and nonspecific mechanisms of action, most conventional chemotherapies result in significant toxicities that limit the effectiveness of treatment and reduce the overall quality of life for cancer patients. Encapsulation of these toxic agents inside lipid-based carrier systems (so-called liposomes) results in passive targeting of the compounds to solid tumors. The preferential delivery of liposomal drugs to solid tumors is mostly due to altered barrier-properties of tumor-associated vessels. This results in both an improved delivery and at the same time a significantly milder toxicity profile. Recently, the specificity of delivery was further increased by attaching monoclonal antibodies or antibody fragments to the surface of liposomes (=immunoliposomes, antibody-linked nanoparticles). Antibody-coated immunoliposomes attach more selectively to antigens expressed on the target cells and they are internalized more efficiently. Furthermore, there is evidence that drug resistance, a major challenge in cancer treatment, may be overcome by such delivery systems. A logical and accessible target, such as EGFR, is overexpressed on a variety of primary human cancer cells and it is involved in signaling pathways that contribute both to tumor initiation and tumor progression. Recently, the investigators have tested immunoliposomes against the epidermal growth factor receptor (EGFR) in a preclinical setting. Based on the preclinical results we have initiated this phase I clinical trial.

Study hypothesis: The investigators hypothesize that anti-EGFR-immunoliposomes selectively deliver cytotoxic compounds to EGFR-overexpressing tumors cells. Specific delivery is supposed to increase efficacy while reducing side-effects of the compound. The primary objective of this phase 1 trial is the determination of the maximum tolerated dose (MTD) for future phase 2 trials of this nanoparticle.

DETAILED DESCRIPTION:
C225-ILS-DOX

This is a phase 1 trial of anti-EGFR-immunoliposomes, an investigative nanoparticle targeted against EGFR-overexpressing tumor cells. The investigators have constructed anti-EGFR immunoliposomes by using Fab' fragments of the chimeric MAb cetuximab (C225, cetuximab, erbitux™, ImClone Systems Corp., NY, USA; Merck KGaA, Darmstadt, Germany), which were covalently conjugated to the liposome membrane. This approach was designed to provide maximal drug delivery to cancer cells via a receptor-targeted and internalizing drug carrier that is stable, non-immunogenic, long-lived with extended blood and tissue residence times and capable of delivering large payloads of diverse types of drugs.

Based on extensive preclinical studies, the investigators decided to perform a first-in-human clinical trial in patients with EGFR-overexpressing solid tumors who have already received all available standard treatments. The therapeutic compound tested in the trial is C225-ILs-dox, a doxorubicin-loaded anti-EGFR-immunoliposome. Doxorubicin is one of the most active agents in many human tumors, and a high percentage of these malignancies do express EGFR. Therefore, the targeting of doxorubicin to EGFR-expressing tumors via the EGFR-specific antibody C225 should enhance the specificity and efficacy of chemotherapy, while the encapsulation of the cytotoxic drug within pegylated liposomes should at the same time decrease its toxicity.

This is a single center, open study. The aim of the trial is the definition of the maximum tolerated dose (MTD) for future phase 2 studies. Secondary endpoints include the overall response rate, the time-to-progression and the assessment of the pharmakokinetic of the compound. The trials follows a canonical 3+3 design and allows an additional recruitment of up to 6 patients on the dose level defined as the MTD. Planned dose levels are as follows:

Level 1 = 5 mg/m2 Level 2 = 10 mg/m2 Level 3 = 20 mg/m2 Level 4 = 30 mg/m2 Level 5 = 40 mg/m2 Level 6 = 50 mg/m2 Level 7 = 60 mg/m2 Level 8 = 70 mg/m2 Level 9 = 80 mg/m2

At each dose level, 3 patients may be enrolled simultaneously. Escalation to the next higher dose will be allowed after patient 3 of a given dose level has received at least one full cycle of therapy if no dose limiting toxicity (DLT) occured at a given dose level. The decision to enter a next dose level will be made by the study team after reviewing all available toxicity data of the previous groups. A DLT is defined as any grade 4 toxicity, any grade 3 toxicity lasting more than one week or/and febrile neutropenia grade 3 (defined as neutrophils < 1.0 x 10e9/l and fever > 38.5 °C). Nausea, vomiting, anorexia, and alopecia (grade 2) will be excluded as dose limiting toxicities. Similarly, adverse events that are clearly related to the primary tumor, such as progression of disease will not be considered as DLTs. In addition, preexisting toxicities must be taken into account when defining and analyzing DLTs.

Patients will be treated until disease progression but for a maximum of 6 cycles. Patients having completed the treatment phase (24 weeks) and showing complete or partial response as well as stable disease will enter the observation phase of the study. This phase will end 12 months after the last patient has been included. At any time during treatment phase or observation phase, patients with signs of disease progression according to RECIST criteria for reporting results of cancer treatment or having discontinued treatment due to unacceptable toxicity will go off study and be treated at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven locally advanced or metastatic solid tumor.
2. ECOG Performance ≤ 2.
3. No additional standard therapy available for the patient.
4. EGFR overexpression (according to DAKO EGFR pharmDx - Test) determined in the most recently evaluable tumor tissue.
5. No concomitant anti-tumor therapy (steroids are permitted - in breast cancer and prostate cancer, steroid dose needs to remain stable during the study period).
6. At least four weeks since termination of any previous anti-tumor treatment (6 weeks in the case of nitrosoureas or mitomycin C).
7. In patients with previous anthracycline exposure, a normal echocardiogram (LVEF > 50%) is required.
8. Age ≥ 18.
9. Male or female.
10. Female and male patients of reproductive age must be using effective contraception.
11. Willing and able to sign an informed consent prior to participation in the study and to comply with the protocol for the duration of the study.

Exclusion Criteria:

1. Pregnancy and/or breastfeeding.
2. Patients with the following laboratory values

   * neutrophils < 1.5 x 109/L
   * platelets < 100 x 109/L
   * serum creatine > 3.0 x upper normal limit
   * ALAT, ASAT > 3.0 x upper normal limit (5.0 x in patients with liver metastases as the only likely cause of enzyme alteration)
   * alkaline phosphatase > 3.0 x upper normal limit (5.0 x in patients with liver or bone metastases as the only likely cause of enzyme alteration)
   * bilirubin > 3.0 x upper normal limit
3. Participation in any investigational drug study within 4 weeks preceding treatment start.
4. Patients with clinically significant and uncontrolled renal- or hepatic disease.
5. Clinically significant cardiac disease: congestive heart failure (New York Heart Association class III or IV); symptomatic coronary artery disease; cardiac arrhythmia not well controlled with medication; myocardial infarction within the last 12 months.
6. Any serious underlying medical condition (at the judgement of the investigator) which could impair the ability of the patient to participate in the trial (e.g. active autoimmune disease, uncontrolled diabetes, etc.).
7. Any concomitant drugs contraindicated when administering Erbitux™ or Caelyx™ according to the Swissmedic-approved product information.
8. A cumulative doxorubicin dose of > 300 mg/m2 BSA (or cardiotoxic anthracycline-equivalent).
9. Patients with a history of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant and precluding informed consent or interfering with compliance.
10. Brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Determination of the maximum tolerated dose (MTD) | after completion of the 1st cycle (day 28)
  The MTD is defined through the occurrence of two dose limiting toxicities (DLTs) at a specific dose level. DLT are defined as any grade 4 toxicity, any grade 3 toxicity lasting more than one week or/and febrile neutropenia grade 3 (defined as neutrophils < 1.0 x 10e9/l and fever > 38.5 °C). Nausea, vomiting, anorexia, and alopecia (grade 2) will be excluded as dose limiting toxicities. Similarly, adverse events that are clearly related to the primary tumor, such as progression of disease will not be considered as DLTs.

SECONDARY OUTCOMES:
CT scans for efficacy | every 2 months for 6 months and then every 3 months for a total of one year

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Mamot, MD, Principal Investigator — Cantonal Hospital of Aarau, Switzerland
Locations (1):
- University Hospital, Basel, Basel, Switzerland

REFERENCES:
- [Background] Mamot C, Drummond DC, Greiser U, Hong K, Kirpotin DB, Marks JD, Park JW. Epidermal growth factor receptor (EGFR)-targeted immunoliposomes mediate specific and efficient drug delivery to EGFR- and EGFRvIII-overexpressing tumor cells. Cancer Res. 2003 Jun 15;63(12):3154-61. PMID 12810643
- [Background] Mamot C, Drummond DC, Noble CO, Kallab V, Guo Z, Hong K, Kirpotin DB, Park JW. Epidermal growth factor receptor-targeted immunoliposomes significantly enhance the efficacy of multiple anticancer drugs in vivo. Cancer Res. 2005 Dec 15;65(24):11631-8. doi: 10.1158/0008-5472.CAN-05-1093. PMID 16357174
- [Derived] Mamot C, Ritschard R, Wicki A, Stehle G, Dieterle T, Bubendorf L, Hilker C, Deuster S, Herrmann R, Rochlitz C. Tolerability, safety, pharmacokinetics, and efficacy of doxorubicin-loaded anti-EGFR immunoliposomes in advanced solid tumours: a phase 1 dose-escalation study. Lancet Oncol. 2012 Dec;13(12):1234-41. doi: 10.1016/S1470-2045(12)70476-X. Epub 2012 Nov 13. PMID 23153506